CLINICAL TRIAL: NCT05909748
Title: First in Human Study of the GEMINUS Transcatheter Aortic Valve Implantation System in Patients With Severe Symptomatic Aortic Stenosis
Brief Title: FIH Study of the GEMINUS TAVI System in Patients With Severe Symptomatic Aortic Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Valve Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMINUS-001
Record Dates: First submitted 2023-05-30; First posted 2023-06-18 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-03

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- GEMINUS Transcatheter Aortic Valve Implantation system (Experimental): Clinical follow up for all patients will be performed at 30 days, 6 months, 1, 2, 3, 4 and 5 years post-implantation
  Interventions: Device: GEMINUS Transcatheter Aortic Valve Implantation system

INTERVENTIONS:
Device: GEMINUS Transcatheter Aortic Valve Implantation system — Implantation of the GEMINUS Transcatheter Aortic Valve Implantation system
  Other Names: GEMINUS TAVI system

SUMMARY:
The main objective of this study is to evaluate the feasibility and safety of the GEMINUS system in patients with severe symptomatic aortic stenosis.

This is a prospective, open label, multicentre, single arm, first in human clinical study.

Clinical follow up for all patients will be performed at 30 days, 6 months, 1, 2, 3, 4 and 5 years post-implantation

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patient understands the implications of participating in the study and provides informed consent
3. Patient is willing to comply with specified follow-up evaluation
4. Severe aortic stenosis as per ACC/AHA 2020 guidelines (e.g. AVA ≤ 1.0 cm2 (or AVA index ≤ 0.6cm2/m2)* AND PV ≥ 4 m/sec or mean gradient ≥ 40 mmHg)** as determined by TTE/CT-TAVI

   *May be larger with mixed AS/AR

   **For low flow low gradient AS or paradoxical low flow severe AS must meet ACC/AHA guidelines (table 13 stages of AS in the guideline)
5. Cardiac Symptoms: ≥ NYHA Class II
6. Patient ≥ intermediate surgical risk as assessed by the heart team or ≥75 years old.
7. Aortic annulus diameter ≥22 mm and < 29 mm, assessed by CT TAVI
8. Anatomically suitable for implantation of the GEMINUS device
9. Peripheral vessels (common femoral and iliac arteries) of acceptable size (minimal diameter > 4mm), tortuosity, and calcification to accommodate the 12Fr catheter system.
10. Patients assessed by the heart team to be at high risk for access site related bleeding/vascular complications due to the caliber/ calcification/ atherosclerosis of the iliofemoral vessels.

Exclusion Criteria:

1. Patient not suitable for surgical bailout
2. Congenital uni/bi/quadricuspid valve, or noncalcified aortic valve.
3. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation ≥3+).
4. Active or recent (within 6 months) endocarditis.
5. Active systemic infections.
6. Recent MI (≤ 1 month).
7. Any therapeutic invasive cardiac procedure (except BAV) performed within 30 days of the index procedure.
8. Prosthetic heart valve in any position.
9. Severe (> 3+) mitral, tricuspid or pulmonic regurgitation.
10. Blood dyscrasias as defined: leukopenia (WBC<3000/mm3), acute anemia (Hb <8mg%), thrombocytopenia (platelet count <50,000 cells/mm3), history of bleeding diathesis or coagulopathy.
11. Untreated clinically significant coronary artery disease requiring revascularization.
12. Hemodynamic instability requiring inotropic support or mechanical support devices.
13. Hypertrophic cardiomyopathy with or without obstruction (HCM).
14. Severe ventricular dysfunction with left ventricular ejection fraction (LVEF) <20%.
15. Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
16. Active peptic ulcer or upper GI bleeding within the prior 3 months.
17. Known hypersensitivity or contraindication to heparin, inability to tolerate antiplatelet therapy or sensitivity to contrast media (which cannot be adequately premedicated).
18. Recent (<6 months) cerebrovascular accident (CVA) or transient ischemic attack (TIA).
19. Renal insufficiency (eGFR<30 mL/min) and/or end stage renal disease requiring chronic dialysis.
20. Severe aortic disease, including abdominal aortic or thoracic aneurysm (lumen diameter > 5cm), marked tortuosity, or severe aortic arch atheroma.
21. Life expectancy < 12 months due to non-cardiac co-morbid conditions.
22. Currently participating in an investigational drug or another device study that has not reached its primary endpoint

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Technical success (at exit from procedure room) | immediately after procedure
  Technical success (at exit from procedure room) composite endpoint:
  Freedom from mortality, Successful access, delivery of the device, and retrieval of the delivery System, Correct positioning of a single prosthetic heart valve into the proper anatomical location, Freedom from surgery or intervention related to the device or to a major vascular or access-related, or cardiac structural complication

SECONDARY OUTCOMES:
Device success composite endpoint | 30 days
  Device success composite endpoint: Technical success; Freedom from mortality; Freedom from surgery or intervention related to the device or to a major vascular or access-related or cardiac structural complication; Intended performance of the valve (mean gradient <20 mmHg, peak velocity <3 m/s, Doppler velocity index ≥0.25, and less than moderate aortic regurgitation)
Early safety composite endpoint (VARC 3) | 30 days
  Early safety composite endpoint: Freedom from all-cause mortality; Freedom from all stroke; Freedom from ≥ VARC-3 type 2 bleeding; Freedom from major vascular, access-related, or cardiac structural complication; Freedom from acute kidney injury stage 3 or 4; Freedom from moderate or severe aortic regurgitation; Freedom from new permanent pacemaker due to procedure-related conduction abnormalities; Freedom from surgery or intervention related to the device
Early safety composite endpoint (Modified VARC) | 30 days
  Early safety composite endpoint: Freedom from all-cause mortality; Freedom from all stroke; Freedom from ≥ Modified VARC type 3 bleeding; Freedom from major vascular, access-related, or cardiac structural complication; Freedom from acute kidney injury stage 3 or 4; Freedom from moderate or severe aortic regurgitation; Freedom from new permanent pacemaker due to procedure-related conduction abnormalities; Freedom from surgery or intervention related to the device
Clinical efficacy composite endpoint | 1, 2, 3, 4, 5 years
  Clinical efficacy composite endpoint: Freedom from all-cause mortality; Freedom from all stroke; Freedom from hospitalization for procedure- or valve-related causes; Freedom from KCCQ Overall Summary Score <45 or decline from baseline of >10 point (i.e. Unfavourable Outcome)
All-cause mortality | 30 days, 6 months, 1, 2, 3, 4, 5 years
  All-cause mortality
Disabling stroke | 6 months, 2, 3, 4, 5 years
  Disabling stroke
Any stroke | 30 days, 6 months, 1, 2, 3, 4, 5 years
  Any stroke
Peri-procedural MI (per ARC-2) | within 2 days after procedure
  Peri-procedural MI (per ARC-2).
Repeat hospitalization for procedure or valve related cause | 30 days, 6 months, 1, 2, 3, 4, 5 years
  Repeat hospitalization for procedure or valve related cause
Repeat aortic valve intervention | 30 days, 6 months, 1, 2, 3, 4, 5 years
  Repeat aortic valve intervention
AKI (Stage 3 or 4) | 30 days
  AKI (Stage 3 or 4)
Bleeding ≥ VARC-3 type 2 | 30 days, 6 months, 1, 2, 3, 4, 5 years
  Bleeding ≥ VARC-3 type 2
Bleeding ≥ Modified VARC type 3 | 30 days, 6 months, 1, 2, 3, 4, 5 years
  Bleeding ≥ Modified VARC type 3
KCCQ- Kansas City Cardiomyopathy Questionnaire | 6 months, 1 year
  Kansas City Cardiomyopathy Questionnaire, 0-5 (none- extremily)
Hemodynamic valve performance: Mean pressure gradient | pre-discharge, 30 days, 6 months, 1, 2, 3, 4, 5 years
  Hemodynamic valve performance: Mean pressure gradient
Hemodynamic valve performance: peak velocity | pre-discharge, 30 days, 6 months, 1, 2, 3, 4, 5 years
  Hemodynamic valve performance: peak velocity
Hemodynamic valve performance: aortic valve area | pre-discharge, 30 days, 6 months, 1, 2, 3, 4, 5 years
  Hemodynamic valve performance: aortic valve area
Hemodynamic valve performance: aortic regurgitation | pre-discharge, 30 days, 6 months, 1, 2, 3, 4, 5 years
  Hemodynamic valve performance: aortic regurgitation
Freedom from new permanent pacemaker due to procedure-related conduction abnormalities | 30 days
  Freedom from new permanent pacemaker due to procedure-related conduction abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Ran Kornowski, Prof., Principal Investigator — Rabin Medical Center
Locations (2):
- Israel (2):
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasly Medical Center, Tel Aviv